CLINICAL TRIAL: NCT05212389
Title: Hormonal Sensitivity and Brain Function: Do Oral Contraceptives Distort Serotonergic Brain Signaling?
Brief Title: The Pill Project - Oral Contraceptive and Serotonergic Brain Signaling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibe G Frøkjær, MD, PhD, MD, Adjunct Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-003366-13
Record Dates: First submitted 2021-12-20; First posted 2022-01-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Major Depressive Disorder; Sexual Behavior; Mood Disturbance; Mood Change; Affect Altered; Affect Blunted; Drug Mechanism
Keywords: Oral Contraceptive; Hormone sensitivity; Positron Emission Tomography; Magnetic Resonance Imaging; Functional Magnetic Resonance Imaging; serotonin 4 receptor; 5-HT4 receptor; (11C)SB207145
MeSH Terms: conditions — Depressive Disorder, Major; Sexual Behavior | interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Intervention Model Description: Single-blinded placebo-controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femicept (Active Comparator): 3x28 days of treatment with Femicept. Each cycle consists of 21 days of active pill (Femicept) and 7 days of placebo pill.
  Interventions: Drug: Femicept
- Placebo (Placebo Comparator): 3x28 days of treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Femicept — 150 μg levonorgestrel +30 μg ethinylestradiol
  Other Names: Combined oral contraceptive
  Arms: Femicept
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Large register based work has shown that starting on oral contraceptives (OCs) is associated with an increased risk of developing depressive episodes. It is not known why this is, but changes in the serotonergic brain system might play a role. Intriguingly, in cross-sectional work, the investigators have demonstrated a lower level of the serotonin 4 receptor globally in the brain of healthy women using oral contraceptives compared to non-users. The order of magnitude of this difference is comparable to what has been observed in depressed individuals relative to healthy controls. In this study, the investigators will apply a longitudinal design to determine if starting on oral contraceptives induces a reduction in the serotonin 4 receptor in healthy women and whether such changes are related to potential changes in measures of cognition as well as mood/affect and sexual desire.

The study is a single-blind randomized placebo-controlled trial with a 3-month intervention paradigm of either Femicept (2nd generation combined oral contraceptive) or placebo. The investigators will include participants until 20 women have completed the study in each arm. Participants will go through an investigational program, including PET and MR brain scans and neuropsychological testing, before starting on the treatment and again during the third pill cycle. To capture changes in mood/ and sexual desire, the participants will complete daily questionnaires during the baseline menstrual cycle and during third pill cycle.

A linear latent variable model will be used to evaluate if OC use induces changes in the serotonin 4 receptor level and such changes will be correlated to changes in secondary outcomes (i.e., cognitive and psychometric measures).

DETAILED DESCRIPTION:
Background:

More than 100 million women worldwide use combined oral contraceptives (OCs), i.e. the most common types that combine estrogen and gestagen. Register-based epidemiological work has recently shown that starting on hormonal contraceptives is associated with an increased risk of developing a depressive episode, and apparently this includes the most severe cases that involve suicide. In addition, the use of OCs has also been linked to reduced sexual desire and interest, one of the common symptoms in depressive disorder. It is unknown why OCs can trigger a depressive episode, at least in a subgroup of women, or how this subgroup at high-risk may be identified in advance.

OCs act by suppressing the hypothalamic-pituitary-gonadal hormonal axis, which drives the reproductive system, resulting in downregulated sex hormones. Such changes in sex-steroid milieu shape human brain biology and function including serotonergic neurotransmission, which is key in maintaining mental health, including regulation of sexual desire. Preliminary and independent data from the Center for Integrated Molecular Brain Imaging (Cimbi) database, strongly suggest that healthy women who use OCs differ in terms of serotonergic brain architecture. In particular when using a potential marker of brain serotonergic function, the investigators have in a cross-sectional study shown, that OC users display lower serotonin 4 receptor (5-HT4R) brain binding relative to non-users. This difference is remarkably large and comparable to what is seen in depressed individuals compared to in healthy controls and to the effects provoked by pharmacological tools as traditional antidepressant drugs (SSRI). The 5-HT4R is relevant in the context of depression, since rodent work points to a fast-acting antidepressant- and anxiolytic-like effect of 5-HT4R stimulation and also, notably, 5-HT4R activation is implicated in behavioral and neurogenic effects of SSRIs. Therefore, a lowered 5HT4R agonism capacity in OC users would offer a plausible explanation for why OC use may provoke depressive symptoms.

The initial cross-sectional observation of a difference in 5-HT4R binding between OC users and non-users warrants replication and validation in an independent dataset and in a study design where causality can be inferred. With this study, the investigators apply longitudinal study design to determine if OC use versus placebo cause changes in 5-HT4R brain binding and if such changes map onto relevant signatures of brain functions and mental states, including sexual desire. The investigators anticipate that this work will substantially advance the understanding of how changes in sex-hormone milieu increase susceptibility for manifest depressive episodes and ideally provide novel preventive and therapeutic opportunities.

Study design:

The investigators will conduct a single-blind randomized placebo-controlled trial with a 3-month intervention paradigm of either OC or placebo. The investigators will include up to 50 healthy women (until 20 women have completed in each arm) at 18-22 years of age. The participants will be allocated to receive a 2nd generation OC (Femicept) or placebo for three pill cycles of 28 days. The participants will undergo an investigational program at baseline (before treatment allocation) and at follow-up (at a specific time in the third pill cycle dependent on treatment arm). The programs consist of 11C-SB207145 PET and MRI/fMRI scan of the brain, neuropsychological testing, collection of blood and saliva samples, completion of questionnaires regarding various trait- and state-related measures including a month at baseline and follow-up of daily questionnaires measuring psychometrics of mood/affect, sexual desire and sleep quality. The participants will be instructed to contact us by e-mail every time they have their first cycle day, i.e. first day of bleeding, during the study, which will be used to estimate menstrual cycle phases.

Randomization:

Participants will be randomized in random block sizes to either Femicept or placebo. The randomization will be carried out by an administrative staff member at Neurobiology Research Unit (Rigshospitalet, Denmark), who will not otherwise be involved in the study or enrollment. The sequence generation will be created via the online service, Sealed EnvelopeTM (www.sealedenvelope.com). Region Hovedstadens Apotek will carry out allocation concealment by sequentially numbered containers. Enrollment and intervention assignment will be carried out by the clinical investigators. The assignment to active or placebo treatment will happen after the baseline assessment. The investigators will be unblinded after a certain time after allocation so they will be able to plan the follow-up investigational program. To evaluate the efficacy of blinding, participants will be asked which group they believed they belonged to prior to unblinding.

Intervention:

Femicept (CampusPharma) is a monophasic 2nd generation combined OC, the recommended type of combined OC due to the lower thromboembolic risk and it is the most used combined OC in Denmark (www.medstat.dk). One packet consists of 21 active pills, containing 150 micrograms levonorgestrel and 30 microgram ethinylestradiol. One pill is taken every day approximately at the same time of the day (with no more than 12 hours variation) for 21 days. Normally, this will be followed by 7 days off the pill before starting on a new pill cycle, however, to decrease complexity and to increase compliance and the timing of pill cycles, a 7-day regime with placebo pills will be added, during which participants will experience withdrawal bleeding. The placebo pill cycle treatment constitutes 28 days with a daily placebo pill.

Evaluation of compliance:

Pill count will be carried out at every pill cycle and plasma estradiol and progesterone will be measured during pill cycle day 18-28 to capture non-compliance based on non-suppressed endogenous ovarian hormone levels indicating if ovulation had occurred. If the participants have missed more than two pills during a pill cycle or if plasma sex steroid levels indicate non-compliance during a pill cycle, it is allowed to extend the treatment with one or two more pill cycles before follow-up, hence, for some participants the intervention may last 4-5 months.

Statistical analysis plan:

The investigators will use linear latent variable models on log-transformed 5-HT4R binding potentials to estimate the multiplicative group effect of OC use (i.e., the percentage change from baseline in 5-HT4R binding potentials) in the regions of interest (neocortex, neostriatum, and the hippocampus) and compare it between the groups. The log-transformed binding potentials will be adjusted for the injected tracer mass per kg body weight. The investigators will compute model diagnostics by using score tests to detect model misspecifications and add parameters until no misspecification can be detected.

Correlation analyses will be used to investigate the association between changes in 5-HT4R binding potentials and secondary outcome measures; affect and sexual desire scores, reward fMRI BOLD signals and verbal memory performances. Mediation analysis will be conducted to test the relation between OC-induced changes in 5-HT4R binding potential and the cortisol awakening response (CAR).

Further, in an explorative approach, the investigators will conduct pooled analyses of baseline data (both OC and placebo group) and potential coupling between baseline imaging outcomes and behavioral outcomes will be performed. Also, analyses of psychometric variations potentially mapping onto menstrual cycle phases will be performed.

Sample size calculation:

Calculations based on intra-subject variability of the 5-HT4R binding on 16 subjects with scan-rescan show that a group size of 20 is required to detect 8-11% difference in 5-HT4R BPND in the region of interest (neostriatum, neocortex, and hippocampus) between OC- and placebo group from baseline to follow-up with a power of 0.8 and a significance level of 0.05 (two-sided). This is equivalent to the effect size seen in the cross-sectional finding for these regions. For the primary analyses, only participants with 5-HT4R follow-up data will be included. Missing data as well as dropouts will be reported in the relevant publications. Dropouts with baseline data can be included in the explorative pooled analyses of the baseline data.

Hypotheses

Primary hypothesis:

1. OC use reduces neostriatal, neocortical, and hippocampal 5-HT4R brain binding from baseline relative to placebo.

   Secondary hypotheses:
2. OC use induces a reduction in positive affect and day to day positive affect variability possibly in a manner dependent on the magnitude of 5-HT4R binding decrease in OC users.
3. OC use induces mood disturbance and lower day to day mood disturbance variability possibly in a manner dependent on the magnitude of 5-HT4R binding decrease in OC users.
4. OC use induces a reduction in sexual desire and day to day sexual desire variability in a manner dependent on the magnitude of 5-HT4R binding decrease in OC users.
5. OC use reduces brain circuit responses to reward stimuli compared to placebo in ventral striatum in a manner dependent on the magnitude of 5-HT4R binding changes.
6. OC use changes resting state functional connectivity brain networks compared to placebo.
7. OC use results in reduced gray matter volumes of the hippocampus.
8. OC use changes white matter integrity.
9. OC use induces a blunted cortisol awakening response (CAR) possibly in a manner dependent on the magnitude of change in 5-HT4R binding and/or changes in hippocampal volume from baseline.
10. The association between 5-HT4R binding and verbal memory performance is dependent on OC use status, such that lower 5-HT4R binding is associated with worse verbal memory performance in the OC use state in contrast to better performance in non-OC use state.
11. OC use results in a bias in processing of emotional information compared to placebo.
12. OC use reduces sleep quality.
13. Within the OC users, the estradiol and/or allopregnanolone levels are associated with the 5-HT4R level, working memory performance, cortisol dynamics and hippocampal volume.
14. OC use induces changes in gene transcript and/or DNA methylation profiles compared to placebo.
15. OC use increases anxiety in a manner dependent on the magnitude of change in 5-HT4R binding.

Ethical considerations:

* Side effects to the intervention: The side effect of most concern is thromboembolic events. However, this risk is only increased from about 1 to 3 per 10.000 women when using 2nd generation OCs, or even less due to the exclusion of those with thromboembolic risk factors, hence it is considered a relatively small risk and acceptable. Further, the blinding of the treatment also raises an ethical concern regarding the risk of pregnancy; even though participants are unaware if they are on OCs or not, they may behave less carefully in regards to preventing pregnancy. To address this, participants will be thoroughly informed to use protection during intercourse and will be offered condoms for free during the study period.
* Exposure to radioactivity during the PET scans: The total exposure will not exceed 10 mSv equal to 3 years of natural background radiation in Denmark, which should be seen in the light of the new knowledge this study can generate.

The study will be conducted in agreement with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women at 18-22 years of age
* No use of hormonal contraception within the last year
* Having a regular menstrual cycle of approximately 28 days, i.e., approximately 28 days between first day of menstrual bleedings.

Exclusion Criteria:

* Current or previous neurological or psychiatric disease, severe somatic disease, or consumption of medical drugs likely to influence the test results
* Non-fluent in Danish or pronounced visual or auditory impairments
* Current or past learning disability
* Current or previous pregnancy
* A wish to become pregnant within the following 6 months
* Participation in experiments with exposure to radioactivity (> 10 mSv) within the last year or significant occupational exposure to radioactivity
* Contraindications for MRI (pacemaker, metal implants, claustrophobia)
* Allergy to the ingredients in the administered drug
* A diagnosis of hypo- or hypertension
* A history of head injury or concussion resulting in loss of consciousness for more than 2 min
* Alcohol abuse
* Drug use other than tobacco and alcohol within the last 30 days
* Cannabis > 50 x lifetime
* Recreational drugs > 10 x lifetime (for each substance)
* Nicotine addiction
* Current psychoactive medication
* Any risk factors for thromboembolic events
* Other contraindications for use of Femicept

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in neostriatal, neocortical, and hippocampal 5-HT4R brain binding from baseline to follow-up measured with Positron Emission Tomography (PET) in active vs. placebo group | 3 months
  Difference in latent variable construct of 5-HT4R level based on a quantification of 5-HT4R binding in primary regions of interest; neocortex, neostriatum, and hippocampus. Change is compared between the OC- and the placebo group.

SECONDARY OUTCOMES:
Change in serial Positive Affect (PA) score derived from daily ratings of the Positive and Negative Affects Schedule (PANAS) questionnaire. | 3 months
  PA score ranges from 10-50 with higher scores representing higher levels of positive affect.
Change in serial Total Mood Disturbance (TMD) scores derived from daily ratings of the Profile of Mood States - Short Form (POMS-SF) questionnaire | 3 months
  TMD score ranges from -30 to 155 with higher scores representing higher levels of mood disturbance.
Change in serial sexual desire scores derived from daily ratings of the Element of Desire Questionnaire (EDQ) | 3 months
  EDQ score ranges from 6-35 with higher scores representing higher sexual desire
Change in the Female Sexual Function Index (FSFI) score | 2 and 3 months
  FSFI score ranges from 2-36 with higher scores representing higher sexual functioning
Change in reward stimulated BOLD signal in ventral striatum measured with fMRI | 3 months
  The blood-oxygen-level-dependent (BOLD) reward signal derived from the brain activity during monetary reward fMRI paradigm
Change in BOLD signal in resting state functional connectivity brain networks measured with fMRI | 3 months
  The blood-oxygen-level-dependent (BOLD) signal derived from the brain activity during resting state.
Change in hippocampal volume | 3 months
  Derived from structural T1 MPRAGE brain MRI
Change in white matter microstructure | 3 months
  Derived from neurite orientation dispersion and density imaging (NODDI) and diffusion tensor imaging (DTI).
Change in CAR | 3 months
  Cortisol Awakening Response (CAR) derived from saliva samples collected during the first hour after awakening
Change in total Verbal Affective Memory Test-24 (VAMT-24) performance | 3 months
  Derived from immediate, short-term and delayed recall with a score range of 0-24 with higher scores representing better performance.
Change in affective bias for emotional detection | 3 months
  Affective bias measures is derived from the Intensity Morphing Task as detection time for sad minus detection time for happy averaged across increase and decrease conditions. Range score is -100% (indicating negative bias) to +100% (indicating positive bias).
Change in affective bias for emotion recognition | 3 months
  Affective bias calculated as hit rate for happy minus hit rate for sad in the Emotion Recognition Task. Range score is -100% (indicating negative bias) to +100% (indicating positive bias).
Change in Letter-Number Sequencing task score | 3 months
  Score ranges from 0-21 with higher scores representing better performance.
Change in mean daily sleep quality | 3 months
  Derived from serial daily sleep quality reporting on a scale from 0 (very good) to 3 (very bad) during baseline and follow-up cycles.
Change in Pittsburgh Sleep Quality Index (PSQI) | 3 months
  PSQI ranges from 0-21 with higher scores representing worse sleep quality.
Plasma estradiol | At baseline and after 3 months
  Sampled at baseline and follow-up
Plasma testosterone | At baseline and after 3 months
  Sampled at baseline and follow-up
Plasma progesterone | At baseline and after 3 months
  Sampled at baseline and follow-up
Serum allopregnanolone | At baseline and after 3 months
  Sampled at baseline and follow-up
Gene transcription and methylation profiles | At baseline and after 3 months
  Derived from mRNA and DNA methylation of genes involved in hormonal signaling pathways
Change in General Anxiety Disorder 10 (GAD-10) score | 2 and 3 months
  GAD-10 score ranges from 0-50 with higher scores representing higher level anxiety

OTHER OUTCOMES:
Change in serial Negative Affect (NA) score derived from daily ratings of the Positive and Negative Affect Schedule (PANAS) questionnaire | 3 months
  NA score ranges from 10-50 with higher scores representing higher levels of negative affect
Change in Positive Affect (PA) score derived from the Positive and Negative Affect Schedule (PANAS) questionnaire (regarding "last few weeks") | 2 and 3 months
  PA score ranges from 10-50 with higher scores representing higher levels of positive affect
Change in Negative Affect (NA) score derived from the Positive and Negative Affect Schedule (PANAS) questionnaire (regarding "last few weeks") | 2 and 3 months
  NA score ranges from 10-50 with higher scores representing higher levels of negative affect
Change in self-reported mental distress scores | 2 and 3 months
  A composite measure derived from Perceived Stress Scale (score range: 0-40, higher score indicating more perceived stress), Snaith-Hamilton Pleasure Scale (score range: 0-14, higher score indicating higher level of anhedonia), Beck Depression Inventory-II (score range: 0-63, higher score indicating more severe depressive symptoms), WHO-5 Well-being index (score range: 0-25, higher score representing higher quality of life), Ruminative Responses Scale (score range: 22-88, higher score indicating higher level of ruminative symptoms), and state-related questionnaires from the State Trait Anxiety Inventory (score range: 20-80, higher score indicating higher level of anxiety) and the State-Trait Anger Expression Inventory 2 (score range: 15-60, higher score indicating higher level of anger)
Change in the 17-item Hamilton Depression Rating Scale (HDRS-17) score | 3 months
  HDRS-17 score ranges from 0-54 with higher scores representing higher level of depressive symptoms
Change in mean hours slept | 3 months
  Derived from serial daily reporting of hours slept during baseline and follow-up cycles
Change in number of nights with trouble sleeping due to 1) difficulty falling a sleep or 2) wakening in the night or early morning | 3 months
  Derived from serial daily reporting about trouble sleeping during baseline and follow-up cycles
Change in visuospatial memory test performance | 3 months
  Derived from immediate, short-term and delayed recall in a Complex Figure Test (CFT) (Taylor CTF will be used at baseline and Reys CTF at follow-up to avoid learning effects). Score ranges from 0-36 with higher scores representing better performance.
Change in Symbol Digit Modalities Test (SDMT) score | 3 months
  Derived from change in number of correct guesses with score ranges from 0-110 with higher scores representing better performance.
Change in Trail Making Test (TMT) Part A and B performance | 3 months
  Derived from time spent with short time representing better performance.
Change in Intra-Extra Dimensional (IED) performance | 3 months
  Derived from Extra Dimensional Set Errors and latency in Intra-Extra Dimensional Set Shifting
Change in Simple Reaction Time (SRT) task | 3 months
  Derived from time spent in trials with shorter time representing better performance.
Color Word Interference Test (CWIT) performance | 3 months
  Derived from test scores in condition 1-4 in D-KEFS Color Word Interference Test (CWIT). The test scores is calculated based on the time spent + corrected errors and uncorrected errors. Shorter time represents better performance.
Verbal Fluency (VF) performance | 3 months
  Derived from test scores from subcategories ("f", "a", "s", "animals", "boy names", "fruit/furniture") in the Verbal Fluency Task
Change in low-grade inflammation | 3 months
  Change in hsCRP from baseline to follow-up
Change in impulsiveness score derived from Barratt Impulsiveness Scale Version 11 | 3 months
  Score ranges from 30-120 with higher score indicating more impulsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Vibe Frokjaer, MD, PhD, Principal Investigator — Neurobiology Research Unit, Copenhagen University hospital, Rigshospitalet, Denmark
Locations (1):
- Neurobiology Research Unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When the planned analyses from the trial are published, the data will become publicly available. According to the Danish legislation, data will be available only by approval by the Danish Data Protection Agency and with a signed agreement.
Supporting Information: Study Protocol
Time Frame: Data are expected to become available from December 2026.
Access Criteria: Data will be available on reasonable request via an application to the Cimbi database of molecular brain PET in healthy humans. Access can be requested through the procedures outlined here: https://cimbi.dk/index.php/documents/category/3-cimbi-database.